CLINICAL TRIAL: NCT06729398
Title: The Role of Cerebral NIRS in Preventing Brain Injury of Very Low Birth Weight Preterm Infants: a Randomized Controlled Trial
Brief Title: The Role of Cerebral NIRS in Preventing Brain Injury of Very Low Birth Weight Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Lily Rundjan, MD, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 623/UN2.F1/ETIK/2016
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Neonatal Cerebral Leukomalacia; Intracranial Nontraumatic Haemorrhage of Fetus and Newborn; Neonatal Mortality
Keywords: Near Infrared Spectroscopy; Intraventricular hemorrhage; Periventricular leukomalacia; Preterm neonates; Very Low Birth Weight
MeSH Terms: conditions — Leukomalacia, Periventricular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: Yes

ARMS (2):
- NIRS and SafeboosC group (Experimental): NIRS is placed on the frontoparietal once the neonates born in the delivery room until 72 hours. SafeboosC treatment guideline is used to maintain normal value of cerebral rStO2.
  Interventions: Device: NIRS; Other: SafeboosC
- Control group (No Intervention): Standard procedure and monitoring device are used for every participant in the control group.

INTERVENTIONS:
Device: NIRS — NIRS is placed on the frontoparietal once the neonates born in the delivery room until 72 hours
  Arms: NIRS and SafeboosC group
Other: SafeboosC — SafeboosC treatment guideline is used to maintain normal value of cerebral rStO2.
  Arms: NIRS and SafeboosC group

SUMMARY:
This study determines the effectiveness of cerebral Near Infrared Spectroscopy (NIRS) as a monitoring device combined with a SafeboosC treatment guideline in order to prevent brain injury in very low birth weight preterm neonates. Each experimental and control groups consists of at least 30 participants, and only the experimental group uses cerebral NIRS and a treatment guideline.

DETAILED DESCRIPTION:
There are still high number of preterm mortality and morbidity in Indonesia. Preterm infants are susceptible to get brain injury due to hemodynamic changes and loss of cerebral autoregulation. Some studies showed that fluctuated changes of brain blood flow caused intraventricular hemorrhage (IVH), and the decreasing of brain blood flow lead to a hypoxic- ischemic state which had role for periventricular leucomalacia (PVL) formation. These result a long term neurologic deficit outcome such as cerebral palsy and cognitive impairment. The standard measures that mainly performed in the NICU were systemic arterial oxygenation and mean arterial blood pressure. There is not yet routine procedure to measure the brain perfusion and oxygenation in Indonesia.

Cerebral Near Infrared Spectroscopy (NIRS) is an invasive tool that continuously measures brain tissue hemoglobin oxygen saturation (rStO2) and determines cerebral circulation. The mechanism of NIRS is based on the light absorption by the hemoglobin, which the value reflects the ratio of oxygenated hemoglobin concentration to total hemoglobin in the penetrated tissue.

To prevent the permanent neurological damage from hypoxia or hyperoxia events, the investigators use cerebral NIRS combined with SafeboosC (Safeguarding the brain of our smallest children) treatment guidelines. The research programme SafeboosC phase II trial hypothesizes that the burden of hypoxia and hyperoxia can be reduced among preterm. The investigators recruit eligible neonates who are admitted in our neonatal intensive care unit and randomly assign them into 2 groups after a written informed consent was approved by the parents. One group uses cerebral NIRS as a monitoring device and performed a treatment guideline to maintain a normal value of rStO2. The other group receives standard treatment without placement of cerebral NIRS. A routine brain ultrasonography is done in both groups to evaluate brain injury (PVL or IVH).

Significance testing is done by Chi-square or Fisher's exact test as needed.

ELIGIBILITY:
* Inclusion Criteria:

  * Neonates born in dr. Cipto Mangunkusumo Hospital and admitted in the neonatal intensive care unit
  * Gestational age ≤ 32 weeks and/or birth weight ≤ 1500grams
* Exclusion Criteria:

  * Parents refuse to participate
  * Participants who are not able to use cerebral NIRS in the first 3 hours of life
  * Participants with congenital malformation and cerebral complications during delivery
  * Participants who are diagnosed with IVH/PVL in the first 3 hours of life (confirmed with brain ultrasonography examination and assessed by radiology pediatric specialist)

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
72 hours preterm brain injury | 72 hours
  Brain ultrasonography at 72 hours of age is assessed by pediatric radiology specialist. Brain injury is positive when there are intraventricular or periventricular leukomalacia findings in the brain ultrasonography result.

SECONDARY OUTCOMES:
Mortality rates | 28 days
  Very low birth weight related mortality rates

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo General Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Data were confidential. Access were only given if the purposes is clear